CLINICAL TRIAL: NCT06426758
Title: The Morbidity of Graves' Disease and Recurrence Rate of Hyperthyroidism Due to Epstein-Barr Virus Lytic Reactivation
Brief Title: Graves' Disease Induced by Epstein-Barr Virus Lytic Reactivation
Status: Not yet recruiting | Type: Observational
Sponsor: Xiao-Ming Mao (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor-Investigator, Xiao-Ming Mao, Professor, Nanjing Medical University
Organization: Nanjing Medical University (Other)
Other Study IDs: NanjingMU2
Record Dates: First submitted 2024-05-19; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Graves Disease; Graves' Disease in Remission; Epstein-Barr Virus
Keywords: Graves Disease; Relapse of hyperthyroidism; Epstein-Barr virus; Lytic reactivation; Morbidity
MeSH Terms: conditions — Graves Disease; Epstein-Barr Virus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Following DNA isolation with a QIAamp DNA Blood Mini Kit, the number of EBV copies in PBMCs was detected using real-time PCR assay by means of the ISEX variant of the EBV PCR kit. The results are expressed in units of EBV DNA copies/µg of DNA, EBV DNA copies/mL of PBMCs suspension, and EBV DNAcopies/100,000 cells.
  Peripheral blood samples were collected from patients with GD and recurrence of hyperthyroidism.Total RNA was extracted from blood using the conventional TRIzol method. Reverse transcription was performed using PrimeScript RT Reagent Kit with cDNA Eraser for two-step reverse transcription polymerase chain reaction.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Previous studies have proved that the lytic reactivation of latent Epstein-Barr virus (EBV) was significantly associated with the onset of Graves'disease (GD), however, the morbidity of GD and recurrence rate of hyperthyroidism after antithyroid drugs treatment due to lytic reactivation of EBV is not understood. We will recruit patients with newly diagnosed GD and recurrence of hyperthyroidism after antithyroid drugs treatment. In order to confirm lytic reactivation of EBV, the number of EBV DNA copies，mRNA and protein expression of immediate-early, early and late lytic EBV genes，EBV +TRAb+cells will be tested. The proportion of lytic reactivation of EBV in newly diagnosed GD and recurrence of hyperthyroidism was evaluated.

DETAILED DESCRIPTION:
The lytic reactivation of latent EBV play importment roles in development of GD and recurrence rate of hyperthyroidism. The aim of this study is to evaluate the proportion of lytic reactivation of EBV in newly diagnosed GD and recurrence of hyperthyroidism.

All patients satisfied the diagnostic criteria for GD. The diagnotic remission of hyperthyroidism was included of clinical symptoms and elevated FT3 and FT4, the patients who have been received antithyroid drugs (methimazole or propylthiouracil) titration treatment for 18 or more months and of antithyroid drugs titration treatment and withdrawal antithyroid drugs at least 3 months.

The evaluation of lytic reactivation of latent EBV including EBV DNA copies，mRNA and protein expression of immediate-early, early and late lytic genes，and EBV +TRAb+cells. The EBV DNA copies was tested with PCR, mRNA and protein expression of immediate-early, early and late lytic EBV genes were analysed with RT-qPCR or Western blot and EBV +TRAb+cells were evaluated with flow cytometry.

All statistical tests were performed using GraphPad Prism V8.0.

ELIGIBILITY:
Inclusion Criteria:

* The clinical evaluation included patient history, physical examination, and thyroid ultrasonography. Laboratory and diagnostic testing included determination of serum levels of free thyroxine (FT4), T3 ( FT3), thyrotropin (TSH), TPOAb, TGAb, and serum levels of thyrotropin receptor antibody (TRAb).

Exclusion Criteria:

* Patients with subacute thyroiditis, hyperfunctioning thyroid nodules, iodine hyperthyroidism, drug-induced hyperthyroidism, or other causes of hyperthyroidism were also excluded. The exclusion criteria for both patients with GD included diabetes, infectious diseases, other chronic diseases, and cancer.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed GD and recurrence of hyperthyroidism after antithyroid drugs treatment
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-05-30 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
The incidence rate of GD and and recurrence of hyperthyroidism due to lytic reactivation of EBV | 3 years
  The GD patients with high number of EBV DNA copies, EBV +TRAb+cells and overexpression lytic genes are considered as lytic reactivation of EBV

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing Medical University, Nanjing, Jiangsu, China